CLINICAL TRIAL: NCT06253897
Title: BackSOM Study: Qualitative Study in Gastro-enteropancreatic Neuroendocrine Tumors (GEP-NETs) and Acromegaly
Brief Title: A Study to Understand Participant's Experiences in Gastro-enteropancreatic Neuroendocrine Tumors (GEP-NETs) and Acromegaly
Acronym: BackSOM
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52030-460
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor; Acromegaly
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants of this study are adults with GEP-NETs and/or acromegaly who were using the Ipsen lanreotide syringe and have transitioned in the last 6 months to the Pharmathen lanreotide syringe, having received at least two injections using the Pharmathen syringe.

GEP-NETs are abnormal growths that develop in the digestive system, including the stomach, intestines, and pancreas. These tumors arise from special cells called neuroendocrine cells, which are found in these organs and release hormones to regulate various bodily functions. GEP-NETs can be slow-growing, and symptoms may vary depending on their location and size.

Acromegaly is a condition where a person's body produces too much growth hormone. This excess hormone can cause certain body parts, like the hands, feet, and face, to enlarge over time. It typically occurs because of a tumor on the pituitary gland in the brain, which is responsible for regulating hormones. Acromegaly can lead to various health issues if not treated, but medications or surgery can often help manage the condition.

Long-acting somatostatin analogs (LA-SSAs) are indicated for patients with Gastroenteropancreatic neuroendocrine tumors (GEP-NETs) and acromegaly who are not eligible for surgery or when surgery fails to achieve remission.

Data for this study will be collected after the treatment switch from the Ipsen lanreotide syringe to the Pharmathen lanreotide syringe has occurred, using one round of one-to-one qualitative telephone and/or videoconference interviews with patients. Interviews will last 45 minutes and be carried out in the local language of the participant's country.

The main aim of this study is to capture the patient experience of the Ipsen lanreotide syringe and their experience with the Pharmathen lanreotide syringe.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients;
* Reside in one of the following countries: France, Italy, Spain, UK and the USA;
* Self-report having a clinician-confirmed diagnosis of GEP-NET and/or acromegaly;
* Have transitioned from treatment with the Ipsen lanreotide syringe to the Pharmathen lanreotide syringe within the last six months and have received a minimum of two injections with the Pharmathen lanreotide syringe;
* Had received a minimum of two injections with the Ipsen lanreotide syringe;
* Switched from the Ipsen lanreotide syringe to the Pharmathen lanreotide syringe only once;
* Are currently being treated with the Pharmathen lanreotide syringe;
* Are willing to provide written informed consent prior to data collection.

Exclusion Criteria:

* Any comorbid condition or factor that, in the opinion of the participants' recruiter or interviewer, may confound the participant's experience or otherwise interfere with their ability to participate fully in a qualitative interview (e.g., speech impediments);
* Participants who switched from independent-injection with the Ipsen lanreotide syringe to HCP-injection with the Pharmathen lanreotide syringe;
* Participants who switched from HCP-injection with the Ipsen lanreotide syringe to independent-injection with the Pharmathen lanreotide syringe;
* USA participants who independently inject (i.e., injections administered by the patient, a family member or friend) with the Ipsen lanreotide syringe and/or the Pharmathen lanreotide syringe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients with GEP-NETs and/or acromegaly living in France, Italy, Spain, UK and the USA
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Qualitative interview: patients' injection experiences and satisfaction with the Ipsen lanreotide syringe and with the Pharmathen lanreotide syringe; | Up to 6 months after treatment switch
  Interview with a duration of 45 minutes.

SECONDARY OUTCOMES:
Qualitative interview: patients' understanding of the reasons for the switch from the Ipsen lanreotide syringe to the Pharmathen lanreotide syringe | Up to 6 months after treatment switch
  Interview with a duration of 45 minutes.
Qualitative interview: patients' perceptions of the Pharmathen lanreotide syringe and of the previous Ipsen lanreotide syringe | Up to 6 months after treatment switch
  Interview with a duration of 45 minutes.
Qualitative interview: patients' preference for the Ipsen lanreotide syringe versus the Pharmathen lanreotide syringe | Up to 6 months after treatment switch
  Interview with a duration of 45 minutes.
Qualitative interview: experiences that are unique to patients who independently inject | Up to 6 months after treatment switch
  Interview with a duration of 45 minutes.
Qualitative interview: experiences that are unique to patients between disease indications | Up to 6 months after treatment switch
  Interview with a duration of 45 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Pearl IRB, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/